CLINICAL TRIAL: NCT05107180
Title: cl[Nical Study of Succide Among Patient With Psychoactive Substance Use Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebat allah hassan goda, residant doctor, Assiut University
Other Study IDs: succide among drug addict
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Drug Screening Assays, Antitumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: drug screen — urine sample

SUMMARY:
detect risk of suicide among patient with substance use disorder

DETAILED DESCRIPTION:
Substance use disorder (or drug addiction) is a neuropsychiatric disorder characterized by recurring desire to continue taking the drug despite harmful consequences. Substance use disorders are a major risk factor for suicide Suicide is a leading cause of premature death in young adults. Data from the World Health Organization indicate that the rate of completed suicide for the world's population is 16 per 100,000 inhabitants, which means that each year more than a million people in the world commit suicide. Suicide attempts are five to twenty times more common than the completed suicide.Based on the data from the research community, approximately 5% of adults attempts suicide at least once in their lifetime .

Mental health problems are the most common and best explored risk factor associated suicidal ideas, suicide attempts and completed suicide. About 90% of all people who commit suicide met the diagnostic criteria for one or more psychiatric disorders . People who use alcohol and/or drugs or are dependent on them, attempting suicide nearly six times more often than people who do not use these substances. The rate of completed suicide among addicts is 2 to 3 times higher than among the males who are not addictst, while in a few cases the manner in which the suicide is attempted is not directly related to drugs . Although there is a correlation between the disorder caused by the use of substances and suicidal behavior, a large number of addicts will never attempt suicide. It is therefore important to identify those individuals with the disorder caused by the use of substances that may be at higher risk for suicide .

Many risk factors for suicide in the general population also apply to drug addicts. The older drug addicts are at higher risk for attempts and suicides than younger addicts Another very important fact when it comes to suicide attempts is the drug used. It is known that heroin and sedatives are substances with which suicide attempts suicide are most often made, while other drugs are less characteristic .

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling diagnostic criteria of substance use disorder

  1. social impairment
  2. impaired control
  3. risky use
  4. pharmacological indicators (tolerance and withdrawal).

Exclusion Criteria:

* Patient with other psychatric disorders ex schizophrenia, mood disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient with substance use disorder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Prevelance of suicide and suicide tendancy in patients with substance use disorders. | 6 months
  observation and study of prevelance of suicide among patient with substance use disorders
Detect risk factors for suicide and in patients with substance use disorder. | 6 months
  observation of patient

REFERENCES:
- [Background] Yuodelis-Flores C, Ries RK. Addiction and suicide: A review. Am J Addict. 2015 Mar;24(2):98-104. doi: 10.1111/ajad.12185. Epub 2015 Feb 2. PMID 25644860
- [Background] Webster LR. Risk Factors for Opioid-Use Disorder and Overdose. Anesth Analg. 2017 Nov;125(5):1741-1748. doi: 10.1213/ANE.0000000000002496. PMID 29049118